CLINICAL TRIAL: NCT00892268
Title: Acupuncture for the Treatment of Aromatase Inhibitor Associated Joint Pain in Post-Menopausal Breast Cancer Patients
Brief Title: Acupuncture or Medication in Reducing Pain in Postmenopausal Women With Breast Cancer and Joint Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accural
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Leona B. Downey, Arizona Cancer Center at University of Arizona Health Sciences Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000629150; P30CA023074 (NIH); UARIZ-07-0792-04; IRUSANAS0084
Record Dates: First submitted 2009-05-01; First posted 2009-05-04 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2009-05

CONDITIONS: Breast Cancer; Menopausal Symptoms; Pain
Keywords: menopausal symptoms; estrogen receptor-positive breast cancer; progesterone receptor-positive breast cancer; breast cancer; pain
MeSH Terms: conditions — Breast Neoplasms; Pain | interventions — Acupuncture Therapy; Analgesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients undergo acupuncture for 20-30 minutes, on the appropriate pain points on the anterior portion of the body alternating with posterior portion of the body, thrice weekly for 2 weeks and then twice weekly for 3 weeks.
  Interventions: Procedure: acupuncture therapy
- Arm II (Active Comparator): Patients receive standard-of-care analgesics (i.e., NSAIDs, narcotics, acetaminophen, or other) for 5 weeks. Patients not responding to analgesia may cross over to arm I.
  Interventions: Procedure: pain therapy

INTERVENTIONS:
Procedure: acupuncture therapy — Undergo acupuncture
  Arms: Arm I
Procedure: pain therapy — Receive standard care
  Arms: Arm II

SUMMARY:
RATIONALE: Acupuncture may reduce joint pain in postmenopausal women with breast cancer. It is not yet known whether acupuncture is more effective than standard therapy analgesics in decreasing joint pain caused by aromatase inhibitors.

PURPOSE: This randomized phase II trial is studying acupuncture to see how well it works compared with medication in reducing pain in postmenopausal women with breast cancer and joint pain.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the efficacy of acupuncture in reducing pain, defined by improvements in overall WOMAC score at 6 weeks, in post-menopausal women with breast cancer and aromatase inhibitor (AI)-associated arthralgia.

Secondary

* To identify biologic correlates to acupuncture efficacy in this specific syndrome of AI-associated pain.
* To evaluate the efficacy of acupuncture in these patients.

OUTLINE: Patients are randomized to 1 of 2 treatment arms:

* Arm I: Patients undergo acupuncture for 20-30 minutes, on the appropriate pain points on the anterior portion of the body alternating with posterior portion of the body, thrice weekly for 2 weeks and then twice weekly for 3 weeks.
* Arm II: Patients receive standard-of-care analgesics (i.e., NSAIDs, narcotics, acetaminophen, or other) for 5 weeks. Patients not responding to analgesia may cross over to arm I.

Patients are assessed periodically for improvement in pain, menopausal symptoms, and overall quality of life by the WOMAC, Brief Pain Inventory, and FACT-ES questionnaires.

Blood samples are collected at baseline, 6 weeks, 3 months, and 6 months for biomarker studies of brain-derived neurotrophic factor and serotonin-transporter gene polymorphisms levels by ELISA.

After completion of study therapy, patients are followed at 1 week, 6 weeks, 3 months, and 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer
* Concurrent therapy with anastrozole for the adjuvant treatment of breast cancer
* Must have moderate or worse arthralgia, as defined by a baseline WOMAC pain scale score ≥ 48

  * Patients with other underlying pain syndromes (e.g., osteoarthritis) are eligible, but the arthralgia must have worsened since starting anastrozole
* Hormone receptor-positive disease

PATIENT CHARACTERISTICS:

* Post-menopausal status meeting the following criteria:

  * At least 12 months without spontaneous menstrual bleeding
  * History of bilateral salpingo-oophorectomy with or without hysterectomy
  * Age > 55 with hysterectomy with or without oophorectomy
  * Age < 55 with hysterectomy without oophorectomy or with unknown status, and serum FSH in post-menopausal range within the past 4 weeks
* Not needle phobic
* Patients with a contraindication to NSAIDs (i.e., prior gastrointestinal bleed secondary to NSAIDs or severe renal insufficiency) are eligible, but will be treated with alternative analgesics such as narcotics or acetaminophen

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Concurrent chronic narcotics or NSAIDs allowed, but doses must be stable for ≥ the past month
* Concurrent antidepressant medications allowed, but doses must be stable for ≥ the past 3 months
* At least 6 months since prior acupuncture
* No prior acupuncture for aromatase inhibitor-associated pain syndrome

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Improvement in pain, as defined by the WOMAC global score at 6 weeks

SECONDARY OUTCOMES:
Acupuncture efficacy as defined by bio-correlates, e.g., changes in BDNF and STGP levels
Menopausal symptoms as defined by the FACT-ES

CONTACTS AND LOCATIONS:
Overall Officials: Leona B. Downey, MD, Principal Investigator — University of Arizona